CLINICAL TRIAL: NCT05208619
Title: Comparison of Different Methods for Intra- and Postoperative Pain Therapy in Thoracic Surgery
Acronym: VERITAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bonn (Other)
Collaborators: HELIOS Klinikum Bonn/Rhein-Sieg (Unknown)
Responsible Party: Principal Investigator, Martin Soehle, Vice Head of Department, University Hospital, Bonn
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Veritas
Record Dates: First submitted 2021-12-09; First posted 2022-01-26 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Thoracic Surgery
Keywords: Thoracic surgery; paravertebral block; epidural analgesia; Thoracic anaesthesia
MeSH Terms: interventions — Anesthesia, Conduction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- thoracic epidural analgesia (Active Comparator): A thoracic epidural catheter is placed before induction of general anaesthesia. Sufentanil 10 µg and Ropivacaine are applied via the catheter.
  Interventions: Procedure: Regional anaesthesia
- paravertebral block (Active Comparator): A single-shot paravertebral block (Ropivacaine 0,5%) is placed before induction of general anaesthesia.
  Interventions: Procedure: Regional anaesthesia

INTERVENTIONS:
Procedure: Regional anaesthesia — Patients receive either a thoracic epidural analgesia or paravertebral block as an regional anaesthetic adjunct to general anaesthesia for thoracic surgery

SUMMARY:
The aim of the study is to determine which regional anaesthesiological technique (thoracic epidural analgesia or paravertebral block) is more suitable for thoracic surgery

DETAILED DESCRIPTION:
Thoracic interventions (lung operations) are associated with considerable postoperative pain, whereby an open surgical procedure via a skin incision (thoracotomy) is more painful than a minimally invasive endoscopic intervention (thoracoscopy). In order to reduce pain, a regional anaesthetic is administered during the induction of anaesthesia, which reduces pain both intraoperatively and postoperatively. In thoracic surgery, thoracic epidural analgesia (PDA) and paravertebral block (PVB) are the main regional anaesthesiological measures used, although it is unclear which of the two procedures is superior in terms of efficiency and effectiveness. Particularly intraoperatively, but also to some extent postoperatively, regional anaesthesia alone is usually not sufficient for pain management. Rather, additional systemic (i.e. intravenous) analgesics (especially opioids) are administered. Therefore, the amount of these additionally administered analgesics is a measure of the efficiency of the regional anaesthesia procedure.

ELIGIBILITY:
Inclusion Criteria:

* elective thoracic surgery
* American Society of Anaesthesiologists (ASA) 1-3 status
* written informed consent

Exclusion Criteria:

* pregnancy
* adipositas (bmi > 30)
* cardiac arrhythmia
* coagulation abnormalities
* chronic pain
* opiate abuses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2022-08-09 (Actual); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Opiate consumption | intraoperative
  intraoperative opiate consumption

SECONDARY OUTCOMES:
pain score | from admission to post-anaesthesia care unit (PACU) until discharge from PACU (up to 1 hour after admission)
  Numeric Rating Scale (NRS), ranging from 0 (no pain) to 10 (worst imaginable pain). A higher NRS score indicates a worse outcome.
postoperative pain | up to day 2 after surgery
  cumulative dose of postoperatively given pain medication
anaesthetic depth | intraoperative
  Bispectral Index
intraoperative nociception | intraoperative
  Nociception Level (NOL)
Patient recovery | at day 1 after surgery
  Quality of Recovery Score (QoR-15) ranging from 0-150, with a higher value representing a better outcome
Patient satisfaction | at day 2 after surgery
  Bauer Satisfaction Questionnaire, consisting of 10 questions on anaesthesia-related discomfort (with 3 answer options: No/ Yes, moderate/ Yes, severe) and 5 questions on satisfaction with anaesthesia care (with 4 answer options: very satisfied/ satisfied / dissatisfied/ very dissatisfied)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Dept. of Anaesthesiology and Intensive Care Medicine, University of Bonn, Bonn
  - Helios Klinikum Bonn/Rhein-Sieg, Bonn

IPD SHARING:
Plan to Share IPD: No